CLINICAL TRIAL: NCT05309447
Title: MuscLSS: Effect of Muscle Fatigue on Spinal Imbalance and Motion in Lumbar Spinal Stenosis: Single Center Observational Pilot Study
Brief Title: Effect of Muscle Fatigue on Spinal Imbalance and Motion in Lumbar Spinal Stenosis
Acronym: MuscLSS
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-02012; mu22Netzer2
Record Dates: First submitted 2022-03-22; First posted 2022-04-04 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Symptomatic Lumbar spinal stenosis (sLSS); Spinal motion; Spinal loading; Spinal imbalance; Paraspinal muscle fatigue; Muscle degeneration; EOS medical imaging
MeSH Terms: conditions — Spinal Stenosis | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with sLSS: Patients with Symptomatic Lumbar Spinal Stenosis (n=10)
  Interventions: Other: data collection
- Young Controls: Young healthy control subjects (n=10)
  Interventions: Other: data collection
- Age-Matched Controls: Age-matched healthy control subjects (n=10)
  Interventions: Other: data collection

INTERVENTIONS:
Other: data collection — The study entails the collection of clinical, functional, radiological, and biomechanical data.

SUMMARY:
This study assesses spinal imbalance and motion in patients with sLSS and elicits fatigue via back exercises and compares spinal imbalance and motion before and after the fatigue exercise and compares these to healthy controls, allowing to associate sLSS-specific motion patterns to paraspinal muscle fatigue.

DETAILED DESCRIPTION:
Symptomatic lumbar spinal stenosis (sLSS) is a common syndrome affecting the human spine characterized by age related degeneration of the lumbar discs and facet joints resulting in pain, limited function and compromised quality of life. In a healthy spine, global and local spinal loads during static posture and dynamic motion will have minimal effects on the spinal canal. However, spinal loads altered by the presence of sLSS may result in further narrowing of the spinal canal and compression of the neural elements or in overloading of the already degenerated lumbar segments possibly eliciting typical pain symptoms. This study assesses spinal imbalance and motion in patients with sLSS and elicits fatigue via back exercises and compares spinal imbalance and motion before and after the fatigue exercise and compares these to healthy controls, allowing to associate sLSS-specific motion patterns to paraspinal muscle fatigue. Additional data generated using magnetic resonance tomography allows detecting and assessing differences in muscle degeneration between sLSS patients and healthy controls. Radiological images from the spine in upright position using EOS, a specialized low-dose x-ray unit will be obtained to allow the calculation of the actual clinical global and local spinal imbalance. Furthermore, this study investigates the outcome of the decompression surgery during a second study visit scheduled 1 year postoperatively. The data obtained here are pilot data that will be critical for designing a larger clinical trial and produce important information for adapting musculoskeletal spine models to simulate spinal imbalance and motion and further defining meaningful outcome parameters.

ELIGIBILITY:
Inclusion Criteria:for patients with sLSS

* age > 30 years
* BMI < 35kg/m2
* diagnosed symptomatic lumbar spinal stenosis
* clinical symptoms for at least 6 months
* intermittent neurogenic claudication with limitations of their walking ability due to symptoms in the lower back and or in one or both legs
* unsuccessful conservative treatment
* confirmation of the LSS through MRI
* Inclusion criteria for age-matched healthy control subjects
* age > 30 years
* BMI < 35kg/m2
* Inclusion criteria for young healthy control subjects
* 18 years ≤ age ≤ 30 years
* BMI < 35kg/m2

Exclusion Criteria:for patients with sLSS

* inability to provide informed consent
* previous spine surgery
* use of walking aids
* other neurologic disorders affecting gait
* MRI incompatibility
* Exclusion criteria for age-matched healthy control subjects
* inability to provide informed consent
* previous spine surgery
* history of claudications
* use of walking aids
* other neurological or orthopaedic conditions that may affect gait
* MRI incompatibility
* Exclusion criteria for young healthy control subjects
* inability to provide informed consent
* previous back injury; previous spine surgery
* use of walking aids
* current injury of any kind

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with sLSS will be recruited at the Department of Spine Surgery at the University Hospital Basel.
  Healthy participants will be recruited via advertisement on the institutional website and the University of Basel marketplace.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-11-11 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Global spinal imbalance assessed using motion capture | approximate duration: 30 minutes at baseline and at 1 year after decompression surgery for patients with sLSS
  Global spinal imbalance calculated from markers placed on specific anatomical landmarks: electromyographic (EMG) electrode placement bilaterally on the multifidus, erector spinae (longissimus), erector spinae (iliocostalis), transversus abdominis, gluteus medius, vastus medialis, tibialis anterior and gastrocnemius medialis muscles. The curvature of the lumbar region during natural stance, natural seated posture, maximum trunk flexion, maximum trunk extension and during walking will be computed from the marker data. A cubic polynomial function will be fit to the marker positions in each time frame, approximating an S-shaped spine curvature with thoracic kyphosis and lumbar lordosis curves and the curvature of the lumbar spine will be computed for each task.

SECONDARY OUTCOMES:
Global spinal imbalance assessed using EOS (upright standing sagittal plane EOS images of the full body including entire spine and pelvis) | approximate duration: 10 minutes at baseline and at 1 year after decompression surgery for patients with sLSS
  Static global and local spinal imbalance will be assessed on the EOS images as the C7 plumb line (C7PL), sagittal vertical axis (SVA) and spinosacral angle (SSA). The discrepancy between SSA and SVA are a sign of the prevalence of static compensation mechanism. The correction angle to a balanced situation will be measured using the full balance integrated method.
Dynamic global spinal imbalance | one time assessment at baseline and at 1 year after decompression surgery for patients with sLSS
  Dynamic spinal imbalance will be assessed as the difference between spinal imbalance during walking compared to standing.
Difference in global spinal imbalance between the fatigued and non-fatigued state | one time assessment at baseline and at 1 year after decompression surgery for patients with sLSS
  The curvature of the lumbar region between the fatigued and non-fatigued state will be computed from the marker data.

OTHER OUTCOMES:
Oswestry disability index (ODI) | one time assessment at baseline and at 1 year after decompression surgery for patients with sLSS
  Disability related to LSS will be assessed using the validated German version of the ODI. The ODI is a standardized questionnaire comprising 10 self-administered parameters quantifying the impact of low back pain on daily life
Quality of life (EQ-5D-5L) | one time assessment at baseline and at 1 year after decompression surgery for patients with sLSS
  Overall health will be assessed using the validated German version of the EQ-5D-5L. The EQ-5D-5L is a generic health-related instrument frequently used in clinical environments to measure quality of life. It comprises 5 questions with Likert response options and a visual analogue scale where patients are asked to rate their overall health from 0 (the worst health imaginable) to 100 (the best health imaginable).
Muscle cross sectional area (MRI)) | one time assessment at baseline and at 1 year after decompression surgery for patients with sLSS (approximate duration: 30 minutes)
  For L1 to L5, the cross-sectional area (CSA) of the abdominal and paraspinal muscles on each side and the CSA of the vertebral body will be measured. The relative CSA (rCSA) and the ratio of LeanCSA to the paraspinal muscle CSA (LeanCSA/CSA) will be calculated for each level and side. This measurement of muscle degeneration (atrophy and fatty infiltration) allows quantifying abdominal and paraspinal muscle degeneration.
Muscle fatigue, assessed as the duration of the fatigue exercise from start until termination | one time assessment at baseline and at 1 year after decompression surgery for patients with sLSS
  Muscle fatigue will be quantified as the slope of the mean frequency and the change in the signal intensity during the modified Biering-Sørensen test. The starting position is the patient/client adopting a half prone lying on a plinth with the superior edge of the iliac crest at the edge of the plinth and the arms crossed over the chest.
  The lower limbs are strategically stabilized with straps. The patient/client is asked to maintains the upper body in a horizontal position and the timer is started.
  The test ends if the patient/client can maintain the said position for 4 minutes (240 seconds) or can no longer maintain the set position before 4 minutes elapses. The stop time is recorded.
Fatigue exercise duration | one time assessment at baseline and at 1 year after decompression surgery for patients with sLSS
  Fatigue exercise duration will be recorded as the duration from start to end of the fatigue exercise.
Local spinal imbalance | one time assessment at baseline and at 1 year after decompression surgery for patients with sLSS
  Local spinal imbalance will be calculated from the reflective markers positioned on the spinous processes.

CONTACTS AND LOCATIONS:
Overall Officials: Cordula Netzer, PD Dr. med., Principal Investigator — Spine Center, University Hospital Basel
Locations (1):
- Spine Center, University Hospital Basel, Basel, Switzerland

REFERENCES:
- [Derived] Koch D, Nuesch C, Ignasiak D, Scharen S, Ferguson SJ, Mundermann A, Netzer C. Age and activity but not lumbar spinal stenosis and muscle fatigue affect sagittal spinal alignment: A pilot study. Clin Biomech (Bristol). 2025 Jul;127:106577. doi: 10.1016/j.clinbiomech.2025.106577. Epub 2025 Jun 1. PMID 40472708